CLINICAL TRIAL: NCT00609362
Title: The Effect of Glitazone Treatment on Bone Marrow and Bone Marrow Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Bente Langdahl, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2007-223
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-03

CONDITIONS: Change in Bone Mineral Density; Change in Bone Marrow Fat Content
Keywords: BMD; Rosiglitazone; Bone marrow fat
MeSH Terms: interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosiglitazone (Active Comparator): 25 women age 60 to 75 years receiving rosiglitazone 8 mg/day
  Interventions: Drug: Rosiglitazone
- Placebo (Placebo Comparator): 25 women 60 to 75 years of age receiving placebo once a day for 14 weeks
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Rosiglitazone — one tablet of rosiglitazone 8 milligrams per day for 14 weeks
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: Placebo pill — One encapsulated placebo pill a day for 14 weeks
  Arms: Placebo

SUMMARY:
Osteoporosis is a generalised bone disease leading to an increased risk of fractures. The disease is caused partly by environmental and partly by genetic factors. It is well known that the fat content of the bone marrow is increased in osteoporotic patients. Animal studies suggest that stimulation of bone marrow stem cells through the molecule PPARgamma with the drug rosiglitazone converts the stem cells to fat cells instead of bone cells thereby decreasing bone strength. In a single study healthy volunteers were treated with rosiglitazone for 14 weeks and had a decrease in bone mineral density.

In the present study we wish to investigate the effect of this treatment on bone and fat tissue. 25 women above the age of 60 will be treated with rosiglitazone 8 mg/day for 14 weeks and compared with 25 women receiving placebo.

The effect will be evaluated as follows:

1. The effect on bone marrow density will be examined by a bone scan prior to and after treatment and again after 6 and 9 months.
2. The effect on bone turnover will be measured in blood- and urine samples at the same times.
3. The effect on fat distribution will be evaluated by an MRI scan after treatment.
4. The effect on bone marrow cells will be investigated bone marrow sampling immediately after treatment
5. The direct effect on fat will be examined by a biopsy immediately after treatment The study hypothesis is that rosiglitazone treatment decreases bone mineral density and increases bone marrow fat content. The causal molecular mechanisms will be investigated from the bone marrow and fat samples

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women age 60-75 with no rosiglitazone allergy

Exclusion Criteria:

* Osteoporosis
* Diabetes
* Hyperthyroidism, untreated hypothyroidism, hyperparathyroidism
* Treatment with bone active drugs
* Low impact fracture
* Heart disease
* Kidney failure
* Liver failure
* Anaemia
* Ineligibility for MRI-scan
* Cancer within last 5 years

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torben Harsløf, Dr., Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment commenced january 2008 and ended february 2009. Participants were recruited by ads in local papers and called our osteoporosis clinic. 179 called and after a course description 150 were sent information. After having read that 74 paid a visit to the clinic.
Pre-assignment Details: 74 individuals were screened. 17 were screen failures due to exclusion criteria. 57 were randomized.
Period: Overall Study
Arm/Group | Rosiglitazone | Placebo
Started | 29 | 28
Completed | 26 | 27
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 14 | 12 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 65.1 (3.5) | 65.3 (4.3) | 65.2 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percent Change in Bone Mineral Density (BMD) From Baseline to 14 Weeks Between the Rosiglitazone Group and the Placebo Group
Description: Difference in percent change in bone mineral density (BMD) from baseline to 14 weeks between the rosiglitazone group and the placebo group. BMD was assesed using dual x-ray absorptiometry (DXA)
Time Frame: BMD measured at baseline and after 14 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 29 | 28
Percent change from baseline | -1.3 (3.1) | 0.3 (2.9)
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; The minimum number of participants was determined by power calculations to be 44 (22 in each group), assuming a difference in change in BMD of 1.7%, a standard deviation of 2%, a power of 80%, and a level of significance of 5%; Test type: Superiority or Other; p = 0.055, t-test, 2 sided — P-value is un-adjusted. A priori threshold for significance: 0.05

2. Secondary Outcome: Difference in Percent Change in Bone Marrow Fat (Given by a Lipid to Water Ratio) in the Spine.
Description: Bone marrow fat was measured using MRI spectroscopy providing a measure of bone marrow fat as a ratio to bone marrow water, the lipid-water ratio (LWR)
Time Frame: Measured at baseline and after 14 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent change in LWR
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 29 | 28
Percent change in LWR | -13.5 (5.5) | 6.8 (24.4)
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; Test type: Superiority or Other; p = 0.056, t-test, 2 sided

3. Secondary Outcome: Difference in Percent Change in Level of C-terminal Telopeptide (CTx) Between the Rosiglitazone and Placebo Groups
Description: C-terminal telopeptide is a marker of bone resorption. Its levels are measure in plasma using a chemiluminometric method (ECLIA).
Time Frame: At baseline and after 14 weeks of treatment
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 29 | 28
Percent change from baseline | 20.4 (38.6) | -7.1 (24.4)
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

4. Secondary Outcome: Change in Gene Expression in Bone Marrow and Fat Cells
Time Frame: Before and after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Rosiglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 19/26 | 15/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone (N=26) | Placebo (N=27)
Cold (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 6 (7) | 4 (4)
Hypercholesterolemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Tendinitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Edema (Cardiac disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes